CLINICAL TRIAL: NCT03368716
Title: Addressing Healthcare Disparities in Pediatric Obesity Treatment: Development of a Novel, Patient-centered Intervention Targeting Executive Function
Brief Title: Acceptance-based Care for Child Eating and Physical Activity Treatment
Acronym: ACCEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Kaul Pediatric Research Institute of the Alabama Children's Hospital Foundation (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marissa Gowey, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5K12HS023009-04 (AHRQ); 5P30DK079626-12 (NIH); in progress (Other Grant/Funding Number: Kaul Pediatric Research Institute of the Alabama Children's Hospital Foundation)
Record Dates: First submitted 2017-11-29; First posted 2017-12-11 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Obesity; Executive Function; Self-Regulation
Keywords: Pediatric Obesity; Executive Function; Behavioral Intervention; Self-Regulation; Acceptance-Based
MeSH Terms: conditions — Pediatric Obesity; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance-based Behavioral Treatment (Experimental): Family acceptance-based behavioral treatment (ABBT) will be piloted with 16 child-caregiver pairs. At weeks 0 (pre-treatment), 9 (mid-treatment), and 18 (post-treatment), feedback regarding the feasibility and acceptability will be collected from participants through surveys and semi-structured group interviews to refine the family ABBT protocol.
  Interventions: Behavioral: Acceptance-based Behavioral Treatment (ABBT)

INTERVENTIONS:
Behavioral: Acceptance-based Behavioral Treatment (ABBT) — ABBT is rooted in behavioral therapy but also cultivates self-regulation skills including experiential acceptance of potentially uncomfortable internal experiences (e.g., emotions, cravings), mindful awareness of decision making (e.g., mindful eating), and values clarification and behavioral commitment (e.g., practicing daily physical activity to be a contributing member on a sports team). ABBT has been used effectively to help youth and adults manage various medical and psychological problems. Moreover, components of ABBT have been shown to improve child and adult EF including inhibitory control and cognitive flexibility. Recently, ABBT has been integrated with components of standard behavioral treatment of obesity and applied with robust efficacy to weight management in adults.

SUMMARY:
The purpose of this study is to develop and pilot test a new type of patient-centered, family-based treatment for children aged 8-12 with obesity and their caregivers. The treatment will focus specifically on improving children's self-regulation (SR) skills to help them better manage their feelings, behaviors, and thoughts to help them live a healthier lifestyle.

DETAILED DESCRIPTION:
We aim to: (1) To determine the treatment needs of children ages 8-12 with obesity and their families with a focus on understanding cognitive function challenges that are related to self-regulation (using focus groups i.e. FG and feedback sessions i.e. FB). (2) To evaluate the feasibility and acceptability of this novel family-based treatment. (3) Explore potential associations between pediatric cardiovascular (CVD) risk factors and self-regulation in children with and without overweight or obesity. (4) To refine the F-ABT protocol and to maximize participant feasibility, acceptability, safety, and tolerability of F-ABT. (5) To provide pilot, proof-of-concept, and preliminary efficacy data of beneficial effects of F-ABT on SR and BMI in children with SR deficits and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

- Children who: (1) have a BMI ≥ 85th percentile; (2) are ≥8 and ≤12 years old at the beginning of treatment; (3) can read, write, and speak English, along with their caregiver; (4) plan to stay living in the local area during the study period; (5) have a consenting caregiver who can commit to all study procedures and provide reliable travel.

Exclusion Criteria:

- Children who:(1) comorbid developmental/intellectual disability/traumatic brain injury/other identified condition known to substantially impact EF and/or weight management; (2) taking medication that is known to affect weight or appetite, (3) recent infection that may cause confounds of acute inflammation, (4) have an uncorrected visual or hearing impairment that would prohibit completion of cognitive testing, and (5) are unable to use an iPad with appropriate training for cognitive testing. The children without obesity (n=32) will have "normal-range" BMI scores (5th ≤BMI percentile< 85th) but otherwise follow the same inclusion/exclusion criteria.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in child body mass index | Baseline to 4.5 months
  Child height and weight measurements will be converted to zBMI using CDC age and sex specific scales.
Change in child objective executive function | Baseline to 4.5 months
  Performance-based EF will be tested using the NIH Toolbox Cognitive Battery which measures executive function (inhibitory control and cognitive flexibility), attention, episodic memory, language, processing speed, and working memory. T-scores will be used for each domain. Higher t-scores indicate better function.
Change in child subjective executive function | Baseline to 4.5 months
  Subjective EF will be measured using the Behavioral Rating Inventory of Executive Function. The Global Severity Index will be used which is interpreted using T-scores. Higher t-scores indicate better function.
Change in Health-Related Quality of Life | Baseline to 4.5 months
  Sizing Me Up© & Sizing Them Up© are validated obesity-specific self-report and parent-report measures, respectively, of health-related quality of life for children 5-13 years old that measure functioning in a variety of areas (e.g., emotional, physical, teasing/marginalization). The Total Score will be used as the outcome, which is a scaled score ranging from 0-100 with higher scores representing better quality of life.
Cortisol | Baseline to 4.5 months
  ug/dl
Blood pressure | Baseline to 4.5 months
  Systolic over diastolic
Fasting glucose | Baseline to 4.5 months
  mg/dl
Low-density lipoprotein (LDL-C) cholesterol | Baseline to 4.5 months
  mg/dl
High-density lipoprotein (HDL-C) cholesterol | Baseline to 4.5 months
  mg/dl
Triglyceride | Baseline to 4.5 months
  mg/dl
Insulin | Baseline to 4.5 months
  uU/ml
Hemoglobin A1C | Baseline to 4.5 months
  Percentage
Leptin | Baseline to 4.5 months
  ng/mL
Tumor necrosis factor (TNF-a) | Baseline to 4.5 months
  pg/ml
Interleukin (IL-6) | Baseline to 4.5 months
  pg/ml
High-sensitivity reactive protein (hsCRP) | Baseline to 4.5 months
  mg/L

SECONDARY OUTCOMES:
Child body fat percent | Baseline to 4.5 months
  The Tanita SC-240 BIA device has been validated for use with children to assess total body fat to the nearest 0.1%. Total body fat percent will be standardized using age and sex specific CDC conversions.
Waist circumference | Baseline to 4.5 months
  The Gulick II anthropometric tape will be utilized to measure children's waist circumference, which will be converted to national published standardized (z) scores.
Child eating behavior | Baseline to 4.5 months
  The Children's Eating Behaviour Questionnaire is a 35-item parent proxy-report measure of eating behavior producing 8 subscales: responsiveness to food, enjoyment of food, satiety responsiveness, slowness in eating, fussiness, emotional overeating, emotional undereating, desire for drinks. Items are scored on a 5-point Likert scale and the mean score of each subscale is used. Higher scores indicate more eating behaviors in a certain domain.
Dietary behavior | Baseline to 4.5 months
  Child and parent dietary habits will be assessed via self-report throughout the intervention using the online USDA SuperTracker software.
Physical activity behavior | Baseline to 4.5 months
  Child and parent physical activity habits will be assessed via self-report throughout the intervention using the online USDA SuperTracker software.
Mindfulness | Baseline to 4.5 months
  The Child Acceptance and Mindfulness Measure (CAMM) is a 10-item measure of children's awareness and acceptance of their own private events or internal experiences. Items are reverse scored on a 5-point Likert scale. Higher scores correspond to higher levels of mindfulness.
Psychological flexibility | Baseline to 4.5 months
  The Avoidance and Fusion Questionnaire for Youth (AFQ-Y) is a 17-item self-report measure for to assess psychological inflexibility in children. Items are scored on a 5-point Likert scale and summed for a total score ranging between 0-68. Higher scores are indicative of greater psychological inflexibility. The Parental Acceptance and Action Questionnaire (PAAQ) is a 15-item measure that evaluates parents' experiential acceptance and action tendencies in the context of their relationship with their children. The Total score is used which is a sum of all items which are rated on a 7-point Likert scale. Higher scores represent a greater degree of parental experiential avoidance.
Impact of the food environment | Baseline to 4.5 months
  The Children's Power of Food Scale is a 15-item self-report assessment of the psychological impact of living in food-abundant environments. Items are rated on a 5-point Likert scale and summed to create a total score. Higher scores reflect greater responsiveness to the food environment.

OTHER OUTCOMES:
Demographics | Baseline
  Child and caregiver characteristics such as age, sex, race/ethnicity, educational level, family income, and marital status will be assessed via caregiver report at baseline only.
Participant satisfaction - interviews | 9 weeks, 18 weeks
  Semi-structured group interviews will assess caregiver and child experiences with the program.
Participant satisfaction - surveys | 9 weeks, 18 weeks
  Surveys will assess the utility of intervention content, intervention burden and satisfaction, participation barriers, and suggestions for change.
Program feasibility - interviews | 9 weeks, 18 weeks
  Semi-structured group interviews will assess caregiver and child experiences with the program.
Program feasibility - surveys | 9 weeks, 18 weeks
  Surveys will assess the utility of intervention content, intervention burden and satisfaction, participation barriers, and suggestions for change.
Adherence - attendance | 9 weeks, 18 weeks
  The number of sessions attended will be the primary indicator of adherence.
Adherence - self-monitoring | 9 weeks, 18 weeks
  As a secondary measure, we will use the number of days that self-monitoring records were completed. A completed self-monitoring record should have at least 2 meals and the total number of exercise minutes recorded per day.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa A Gowey, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Given the small number of participants involved in various aspects of the pilot study, we currently do not plan to widely share individual participant data to maximize confidentiality. Individual requests will be considered.